CLINICAL TRIAL: NCT01623362
Title: Low-fluoride Acidic Liquid Dentifrice in Non-fluoridated Communities: a Randomized Clinical Trial
Brief Title: Evaluation of a Low Fluoride Dentifrice for Caries Control
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Fabio Correia Sampaio, PhD, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LOWF-UFPB
Record Dates: First submitted 2012-05-18; First posted 2012-06-20 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-05

CONDITIONS: Dental Caries
Keywords: Dentifrices; Dental Caries; Fluorides; Nails; pH
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low-fluoride acidic dentifrice (Experimental)
  Interventions: Other: Low-fluoride acidic dentifrice
- Conventional dentifrice (No Intervention): 1100µgF/g-pH7.0
  Interventions: Other: conventional dentifrice
- neutral pH and low-fluoride dentifrice (Experimental): 550 ppm pH 7
  Interventions: Other: neutral pH and low-fluoride dentifrice

INTERVENTIONS:
Other: Low-fluoride acidic dentifrice — 550 ppm (mg/L) of sodium fluoride in pH 4,5; 12 months , 3 times a day.
  Other Names: G1
  Arms: Low-fluoride acidic dentifrice
Other: conventional dentifrice — 1100 ppm (mg/L) of sodium fluoride, pH 7 , 3 times a day for 12 months
  Other Names: G2
  Arms: Conventional dentifrice
Other: neutral pH and low-fluoride dentifrice — 500 ppm sodium fluoride, pH 7 , 3 times a day for 12 months
  Other Names: G3
  Arms: neutral pH and low-fluoride dentifrice

SUMMARY:
The aim of this randomized clinical trial is to evaluate the effect of pH and fluoride concentration in liquid dentifrices in the control of dental caries in early childhood, in non-fluoridated area. This study also aims to assess the effect of the consistency of liquid dentifrices in the fluoride uptake in the plaque and the fluoride concentration in the toenails, to estimate the fluoride intake from these formulations.

DETAILED DESCRIPTION:
The study was carried out with schoolchildren living in a non-fluoridated area, with (A) or without (I) active caries lesions, were randomly allocated into 3 groups according to the LD used over 12 months: Group 1 (n=39-A/38-I): 550µgF/g-pH4.5, Group 2 (n=33-A/35-I) 1100µgF/g-pH7.0, Group 3 (n=33-A/34-I): 550µgF/g-pH7.0.

ELIGIBILITY:
Inclusion Criteria:

* Age 2 to 4 years;
* Not having participated in any other clinical study within 3 months prior to selection;
* Not having very large carious lesions or dentin sensitivity during the study;
* Signature of informed consent by the parents.

Exclusion Criteria:

* Using orthodontic appliances

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 212 (Actual)
Dates: Start 2010-09; Primary Completion 2011-07 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of the concentration of fluoride incorporated into the biofilm and nails 6 months after initiation of dentifrices use in non-fluoridated communities | 6 months
  Samples of plaque and nails were analysed for fluoride using an ion-specific electrode after diffuusion with hexamethyldisiloxane-facilitated (HMDS)

SECONDARY OUTCOMES:
New caries diagnostic criteria: caries progression/regression in caries-active children and caries progression in caries-inactive children after 12 months according to the type of dentifrice used in non-fluoridated communities | 12 months
  The caries progression/regression of active noncavited and progression of inactive noncavitated was evaluated by the date from the examinations at baseline and after 12 months using Nyvad, Machiulskienec, Baelum,1999: Score 0: Sound/ Score 1: Active caries (intact surface)/Score 2: Active caries (surface discontinuity)/Score 3: Active caries (cavity)/Score 4: Inactive caries(intact surface) /Score 5: Inactive caries (surface discontinuity) /Score 6: Inactive caries(cavity)/Score 7: Filling (sound surface)/Score 8: Filling + active caries/Score 9: Filling + inactive caries

CONTACTS AND LOCATIONS:
Overall Officials: Fábio Sampaio, PhD, Principal Investigator — Paraíba Federal University
Locations (1):
- Paraíba Federal University, João Pessoa, Paraíba, Brazil